CLINICAL TRIAL: NCT01502046
Title: A Double Blind, Randomized, Cross Over, Placebo Controlled Phase 2 Clinical Trial to Asses Neuroprotection by Cannabinoids in Huntington's Disease
Brief Title: Neuroprotection by Cannabinoids in Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SAT-HD; 2010-024227-24 (EudraCT Number)
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease, cannabinoids
MeSH Terms: conditions — Huntington Disease | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental)
  Interventions: Drug: delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) — Sativex 2.7 mg delta-9-tetrahydrocannabinol/2.5 mg cannabidiol Oromucosal Spray. One spray per day, up to a maximum of 12 sprays per day.
  Arms: Sativex
Drug: Placebo — Placebo, One spray per day, up to a maximum of 12 sprays per day.
  Arms: Placebo

SUMMARY:
Huntington's disease (HD) is a progressive neurodegenerative disorder, related to an abnormal expansion of CAG triplets in the huntingtin gene, characterized by motor, cognitive and behavioral abnormalities, without known effective symptomatic treatment and without known disease slowing strategy. The most severe neuropathological lesions observed in HD take place in the striatum, one brain area important in motor control and rich in cannabinoid receptors (CBR). CBR are subdivided in two classes: CB1R are located in neurons and play a role in neuronal function; CB2R in brain are located mostly in microglia and modulate neuroinflammation.

CBR disappear early in the course of HD, before there is a massive drop out of cells in the striatum. Cannabinoid transmission is also an early event in brains of animal models of HD. In R6/2 mice, which carry large CAG expansions and develop an early and severe HD phenotype the suppression of the CB1R gene further accelerate the development of a severe clinical syndrome and the characteristic brain inclusions and abnormalities of synaptic density. R6/2 treated mice treated with cannabinoids improve their clinical phenotype, their brain lesions, the synaptic density and the levels of BNDF, a neurotrophic factor which enhances survival and resistance of striatal neurons.

Preliminary studies of cannabinoids in patients with HD have shown that these compounds are safe in these patients. Those studies, however, did not show efficacy because 1) they were underpowered from the statistical point of view, 2) were performed with isolated pure cannabinoids, instead of the more physiological stimulation with a mixture of compounds, and 3) they did use insensitive clinical parameters instead of sensitive end points, such as pathogenically important biomarkers.

The investigators propose a phase II trial with combination of cannabinoids with evaluation of safety, by the profile of adverse events, and efficacy, according to changes of important biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HD
2. Older than 18 years.
3. Able to understand the study, to attend the study visits and to provide informed consent.
4. Stable baseline medication for at least 6 weeks prior to randomization.
5. Score in the UHDRS-motor from 5 to 50.
6. Good cognitive status (MMSE> 25) at the screening visit, with no evidence of major depression, at the discretion of the attending physician, and no evidence of psychosis.
7. Not consumers of products derived from marijuana.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of drug addition.
3. History of psychosis or with history of suicidal attempt.
4. Patients with diseases of the oral cavity that prevents the safe administration of the drug.
5. Patients in which drug administration is contraindicated according to the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events reported | 8 months
Changes in the UHDRs Score | On week 4 and 12 of each period
  UHDRS scale scores from the following perspectives: motor, cognitive, psychiatric and functional.

SECONDARY OUTCOMES:
Changes in the BDNF levels (Brain-derived Neurotrophic Factor), oxidative stress (due to mitochondrial dysfunction) and proinflammatory cytokines in plasma | Basal and on week 4 and 12 of each period
Changes in the BDNF levels (Brain-derived Neurotrophic Factor), oxidative stress (due to mitochondrial dysfunction) and proinflammatory cytokines in cerebrospinal fluid. | On week 12 of each period

CONTACTS AND LOCATIONS:
Overall Officials: Justo García de Yébenes, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lopez-Sendon Moreno JL, Garcia Caldentey J, Trigo Cubillo P, Ruiz Romero C, Garcia Ribas G, Alonso Arias MA, Garcia de Yebenes MJ, Tolon RM, Galve-Roperh I, Sagredo O, Valdeolivas S, Resel E, Ortega-Gutierrez S, Garcia-Bermejo ML, Fernandez Ruiz J, Guzman M, Garcia de Yebenes Prous J. A double-blind, randomized, cross-over, placebo-controlled, pilot trial with Sativex in Huntington's disease. J Neurol. 2016 Jul;263(7):1390-400. doi: 10.1007/s00415-016-8145-9. Epub 2016 May 9. PMID 27159993